CLINICAL TRIAL: NCT06907212
Title: Human Adipocytes - Transcriptional Network Changes Associated With Obesity
Brief Title: Transcriptional Changes in Isolated Human Adipocytes During Obesity
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: S-20200123
Record Dates: First submitted 2024-12-16; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Obesity, Abdominal; Adiposity
Keywords: Human primary adipocytes; Obesity; Systems-wide biology; Gene regulatory networks
MeSH Terms: conditions — Obesity, Abdominal; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Isolated adipocytes of human adipose tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Male and female participants with various BMI: Both male and female participants will be included, with the goal of creating a cohort in which all levels of BMI are equally present. Adipocytes of the abdominal subcutaneous and visceral adipose tissue depots will be isolated and sequenced to perform linear regression analysis of transcriptional networks across BMI.

SUMMARY:
Adipocytes play an important role in our body through their function as metabolic energy stores in the form of fat deposits, which are stored when metabolic energy is in excess and released when energy levels are low. In severe obesity, adipose tissue grows through the production of more adipocytes from stem cells (hyperplasia) and the increase in the size of existing adipocytes (hypertrophy). This ability of adipocytes, to maintain their functionality during tissue expansion, is critical in determining the development of obesity-related comorbidities. However, not all adipocytes are the same as adipocyte function differs greatly depending on the depot in which they are found. To elucidate the mechanisms underlying adipocyte adaptability, it is necessary to obtain a deep systems biology understanding of how signaling in different types of adipocytes regulates metabolism and function. Currently, this research group is conducting a systems biology analysis of adipocyte plasticity in obesity in mouse models, but adipose tissue biopsies from different depots in humans are lacking and needed to investigate the regulation of adipocyte function and plasticity in humans. Such studies of adipocytes are crucial for the understanding how obesity affects adipose tissue function and leads to comorbidities.

DETAILED DESCRIPTION:
The development of overweight and obesity is associated with major changes in adipose tissue, including structural changes in cell type composition as well as gene expression in individual adipose tissue cell types. The molecular mechanisms underlying these changes are not yet known. The investigators therefore hypothesized that overweight and obesity cause changes in the transcriptional program of adipocytes and this leads to impaired function of adipocytes. This study will use advanced genomic technologies available that can measure the dynamic changes in the transcriptome and genomic landscape of isolated adipocytes from patient biopsies, to better understand which changes in the adipocytes in particular underlie the severe comorbidities that occur with the development of obesity. It is expected that the described project will contribute important knowledge about adipocyte-specific transcriptional programs that play a crucial role in obesity. This and thus may contribute to the knowledge required to develop adapted- and personalized medicines, or new therapeutic approaches to treat obesity and its associated diseases.

Recruitment of 100 subjects will be from patients referred for surgical cholecystectomies, herniotomies or similar operations at Bispebjerg Hospital. The control group will consist of study participants with a BMI ≥ 19 kg/m2 and < 25 kg/m2, and the "case" group will consist of study participants with a BMI ≥ 25 kg/m2. When including subjects, emphasis will be placed on achieving a control group of approximately 25 subjects and a "case" group of approximately 75 subjects with varying degrees of elevated BMI.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* BMI> 19 kg/m2
* Can receive oral and written information and give appropriate consent

Exclusion Criteria:

* Active viral hepatitis, HIV positive
* Autoimmune diseases (i.e. lupus)
* Chronic use of corticosteroids (cortisone)
* Unable to give appropriate consent
* Contraindications for biopsy: bleeding tendency.
* Cancer or other comorbidity with an expected survival time of less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruitment of subjects will be from patients referred for surgical cholecystectomies, herniotomies or similar operations, at Bispebjerg Hospital.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Adipocytes specific signaling | June 2024 - Sept 2025
  RNA sequencing of isolated adipocytes
Gene regulatory networks | June 2024 - Sept 2025
  ATAC sequencing of isolated adipocytes to determine the accessible chromatin regions.

SECONDARY OUTCOMES:
Adipocyte cell size | Sept 2024 - Dec 2024
  Determining the average adipocyte cell size and cell size distribution in both tissue depots.
Standard blood tests | Jan 2025 - Sept 2025
  Analysis of standard blood tests by research diagnostics department of the hospital; including nutritional status (haemoglobin, magnesium, zinc, phosphate, ferritin, iron, albumin. Vitamin D, urea), coagulation (INR, APTT, platelets), blood lipids (total cholesterol, LDL, HDL, triglycerides) and insulin resistance (HOMA-IR, HbA1c, C-peptide, glucose).
Adipokine secretion | Jan 2025 - Sept 2025
  Storage of extra serum and plasma for additional analysis of adipokines such as Adiponectin and Leptin.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Mandrup, PhD, Principal Investigator — s.mandrup@bmb.sdu.dk
Locations (1):
- Bispebjerg hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website of main investigating party — https://www.sdu.dk/en/adiposign